CLINICAL TRIAL: NCT05367869
Title: Impact of Intraoperative Spraying Methylene Blue In Thyroidectomy
Acronym: methylene
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qena Oncology Center (Other Government)
Responsible Party: Principal Investigator, Mohamed Ahmed Orabi, specialist of Surgical Oncology, Qena Oncology Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Qena Oncology Center
Record Dates: First submitted 2022-04-28; First posted 2022-05-10 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Impact of Intraoperative Spraying Methylene Blue In Thyroidectomy
Keywords: methylene blue; spraying; intraoperative; thyroidectomy
MeSH Terms: interventions — Thyroidectomy

STUDY DESIGN:
Intervention Model Description: Impact of Intraoperative Spraying Methylene Blue In Thyroidectomy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative Spraying Methylene Blue In Thyroidectomy (Experimental)
  Interventions: Procedure: Impact of Intraoperative Spraying Methylene Blue In Thyroidectomy

INTERVENTIONS:
Procedure: Impact of Intraoperative Spraying Methylene Blue In Thyroidectomy — General anaesthesia ,supine position with hyperextension to the neck Low collar incision to the neck , incision to the skin and platysma muscle and fascia ,upper and lower flaps are developed ,separation of strap muscles and identification of the thyroid gland after freeing of investing fascia Ligation of the middle thyroid vein and ligation and separation of the superior pedicle away from the external laryngeal nerve At this point of operation and before ligation of inferior pedicle methylene blue 0.05% spraying is applied to the field the amount varies according to size of the thyroid lobe and variation in population and neck size Thyroid gland stained by bluish color , recurrent laryngeal nerve not stained or minimally stained so we can avoid injury to it parathyroid glands get red of the stain after about 3 minutes so we can avoid injury to it thyroid gland lose its stain in about 15 minutes so we can remove any residual and decrease residual tissue or recurrence

SUMMARY:
Impact of Intraoperative Spraying methylene blue In thyroidectomy

DETAILED DESCRIPTION:
General anaesthesia ,supine position with hyperextension to the neck Low collar incision to the neck , incision to the skin and platysma muscle and fascia ,upper and lower flaps are developed ,separation of strap muscles and identification of the thyroid gland after freeing of investing fascia Ligation of the middle thyroid vein and ligation and separation of the superior pedicle away from the external laryngeal nerve At this point of operation and before ligation of inferior pedicle, methylene blue 0.05% spraying is applied to the field the amount varies according to size of the thyroid lobe and variation in population and neck size Thyroid gland stained by bluish color , recurrent laryngeal nerve not stained or minimally stained so we can avoid injury to it parathyroid glands get red of the stain after about 3 minutes so we can avoid injury to it thyroid gland lose its stain in about 15 minutes so we can remove any residual and decrease residual tissue or recurrence

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Age more than 15 years
* All pathologies need surgery eg. (mutinodular goiter, malignancy , thyroid nodule,…..etc
* Total thyroidectomy

Exclusion Criteria:

* Pregnant females
* Previous neck surgery or recurrent thyroid surgery
* Subtotal or partial thyroidectomy
* Age less than 15 years
* Preoperative affection to vocal cord
* Preoperative hypocalcaemia

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Recurrent laryngeal nerve injury | 2 weeks
Parathyroid gland Injuries | 3 months
Intraoperative injury to trachea | 2 weeks
Operative time | 1 day
Presence of residual or recurrence | 3 months

SECONDARY OUTCOMES:
Hoarseness of voice | 3 months
  temporary or permanent (by clinical evaluation and vocal cord examination)
Stridor | 3 months
  temporary or permanent (by clinical evaluation and vocal cord examination)
Hypoparathyroidism | 3 months
  temporary or permanent (level of para thormone hormone )
Hypocalcaemia | 3 months
  temporary or permanent ( level of total and free serum calcium )

CONTACTS AND LOCATIONS:
Overall Officials: Remon Elia Lukas, Specialist Surgical Oncology, Study Director — Qena Oncology Center; Mohamed Taha Mousa, Resident Surgical Oncology, Study Director — Qena Oncology Center; Mina Romany Tawfeek, Specialist General Surgery, Study Director — Qena Oncology Center; Abdullah Atyah Ali, Ass.Lecture General Surgery, Study Director — Qena Oncology Center--Luxor University; Ali Hassan, Resident General Surgery, Study Chair — Qena Oncology Center --Qena University; Mohamed Ahmed Orabi, Specialist Surgical Oncology, Principal Investigator — Qena Oncology Center; Amr M Makky, Specialist Surgical Oncology, Study Director — Qena Oncology Center- Medical Military Academy; Mostafa Sayedd Abd el Rahaman, Resident Surgical Oncology, Study Chair — Qena Oncology Center; Mena Zarief Malaty, Resident General Surgery, Study Chair — Qena Oncology Center--Nag hammady Hospital; Hussein El Lithy, Resident General Surgery, Study Chair — Qena Oncology Center--Qena General Hospital; Abobakr Mohammed, Resident General Surgery, Study Chair — Qena Oncology Center--Qena General Hospital; Mohamed Mahmoud El Zeer, Resident General Surgery, Study Chair — Qena Oncology Center- Sohag University; Mahmoud Rabeea Ahmed, Resident General Surgery, Study Chair — Qena Oncology Center-Aswan University; Mohamed Abouelmagd Salem, Prof. Surgical Oncology, Study Chair — Qena Oncology Center-ٍSouth Egypt Center Institute Assiut University; Mohamed Saeed Ayaty, Ass.Prof. Surgical Oncology, Study Chair — Qena Oncology Center-National Cancer Institute Cairo University; Mohamed H Mahran, Ass.Prof. Surgical Oncology, Study Chair — Qena Oncology Center-ٍSouth Egypt Center Institute Assiut University; Mohamed Hasan Abdel-Aal, Director of QOC, Study Chair — Qena Oncology Center

IPD SHARING:
Plan to Share IPD: Yes
Impact of Intraoperative Spraying methylene blue thyroidectomy
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: about 1year